CLINICAL TRIAL: NCT04783831
Title: Usefulness of Biodegradable Pancreatic Stents for the Prevention of Postoperative Pancreatic Fistula After Cephalic Pancreaticoduodenectomy. Prospective Non-randomized Controlled Clinical Study Comparing Biodegradable vs Non-biodegradable Stents
Brief Title: Biodegradable Pancreatic Stents for the Prevention of Postoperative Pancreatic Fistula After Cephalic Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, David Ferreras, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: ARQUIMEDES
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Fistula; Pancreas Neoplasm; Stent Disintegration; Pancreatic Cancer; Pancreatic Anastomotic Leak
Keywords: pancreaticoduodenectomy; pancreaticojejunostomy; pancreatic stent; pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Biodegradable stent
  Interventions: Device: Biodegradable stent
- Non-biodegradable stent
  Interventions: Device: Biodegradable stent

INTERVENTIONS:
Device: Biodegradable stent — Biodegradable stent (polymeric prostheses) is placed from the pancreatic duct to the jejunum. Duct-to-mucosa end-to-side anastomosis is performed for the pancreaticojejunal anastomosis.

SUMMARY:
Background: postoperative pancreatic fistula (POPF) remains the most important morbidity after pancreaticoduodenectomy (PD). There is no consensual technique for pancreatic reconstruction and many surgeons use a transanastomotic drain. Currently, the stents used are not degradable and they can cause obstruction, stricture and pancreatitis. The use of biodegradable stents that disappear a few months after the intervention could have a role in the prevention of pancreaticojejunostomy complications.

Material and method: A single-center prospective randomized study was planned with patients undergoing PD. A duct-to-mucosa end-to-side anastomosis is performed for the pancreaticojejunal anastomosis and the stent is placed from the pancreatic duct to the jejunum.

The primary outcome of the study is the evaluation of the presence of POPF (drainage fluid amylase value of > 5000 U/L on the first day).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cephalic pancreaticoduodenectomy (Whipple procedure).

Exclusion Criteria:

* Patients with soft pancreas or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cephalic pancreaticoduodenectomy (Whipple procedure).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
POPF | 1 week
  Evaluation of the presence of POPF (drainage fluid amylase value of > 5000 U/L on the first day).

SECONDARY OUTCOMES:
Position and degradation of biodegradable stents | 3 months
  Evaluation of the position and degradation time of the biodegradable stents

CONTACTS AND LOCATIONS:
Locations (1):
- David Ferreras, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No